CLINICAL TRIAL: NCT00305500
Title: Phase III Open Study of High Dose Escitalopram for the Treatment of Obsessive-Compulsive Disorder in Adults
Brief Title: Tolerability and Efficacy of High Dose Escitalopram for the Treatment of Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abarbanel Mental Health Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EscitaHD001
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Escitalopram
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
Objectives: To evaluate tolerability and efficacy of escitalopram treatment in high dose than 20-50 mg/d in out-patients with OCD Type of the study: Open label, prospective study.

Number of patients: 100 patients with OCD

Duration of the study: 18-weeks of active treatment, 8-visits:

Dose titration:

One week of 10mg Four weeks of 20mg After 4 weeks of 20mg treatment- if partial/no response, according to YBOCS score and clinical judgment, dose increase of up to 50mg depending on response, adverse events, patient preference and judgment of the clinician 12 weeks follow up on high dose. Total of 18 weeks of follow-up.

DETAILED DESCRIPTION:
Objectives: To evaluate tolerability and efficacy of escitalopram treatment in doses higher than 20mg (20-50 mg/d) in patients with OCD, non responsive or partially responsive to recommended doses.

Type of the study: Open label, prospective study. Study location: Subjects will be recruited from patients treated in a large clinic specializing in mood disorders and anxiety and OCD.

Backup site: the ABARBANEL mental health center. Number of patients: 100 patients with OCD

Duration of the study: 18-weeks of active treatment, 8-visits:

Dose titration:

One week of 10mg Four weeks of 20mg After 4 weeks of 20mg treatment- if partial/no response, according to YBOCS score and clinical judgment, dose increase of up to 50mg depending on response, adverse events, patient preference and judgment of the clinician 12 weeks follow up on high dose. Total of 18 weeks of follow-up.

Patients

Inclusion Criteria:

1. Men and women over 18 years of age
2. DSM IV-TR criteria for OCD
3. OCD associated with most distress or most interference in the patient's life as judged by the treating physician
4. Yale-Brown Obsessive Compulsive Scale (YBOCS) total score ≥16

Exclusion Criteria:

1. Other primary or co-primary psychiatric disorder which is more distressful for the patient then the OCD, as evaluated by investigator
2. Patients with any history of mania/bipolar disorder
3. Patients using medications which are contraindicated with the use of escitalopram
4. Known contraindication for the use of citalopram or escitalopram.
5. Unable to understand and give informed consent
6. Prominent suicidal ideation (2 points or more in the MADRS "suicidal thoughts" item)
7. Alcohol or substance dependence in the past 6 months
8. Major physical illness
9. a) woman currently pregnant or less then 4 weeks after a childbirth Or b) woman lactating Or c) A woman of childbearing potential not using a medically accepted form of contraception.
10. Liver function abnormality
11. EKG abnormalities

Study Design:

An institutional review board acknowledged by the Israeli Ministry of Health will approve the study. After complete description of the study to the patients, written informed consent will be obtained from patients found eligible and willing to participate. The design will be open-labeled. The study will last for 18 weeks.

Patients will be evaluated by clinical assessment and by various questionnaires (see "rating scales" section). Those who will be diagnosed as having OCD and will fulfill the inclusion and exclusion criteria requirements will start 4 weeks of initial treatment with escitalopram up to 20mg/d. After 4 weeks those patients who will be evaluated as non-responders (reduction of Y-BOCS total score by less than 25%) will continue treatment with higher escitalopram dose.

Dose will be adjusted according to clinical status and the clinician's judgment up to 50mg/d of escitalopram. Patients will be evaluated periodically throughout the study for adverse reactions and psychiatric status by various rating scales as well as a clinical evaluation by the investigator.

Assessments:

1. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Symptom Checklist
2. Montgomery Åsberg Depression Rating Scale (MADRS)
3. The Clinical Global Impression scales (CGI) consist of two sub-scales:

   The Severity of illness (CGI-S) and the Global improvement (CGI-I).
4. A checklist of serotonergic specific adverse drug reactions + dizziness, bleeding and ecchymoses checklist
5. Visual Analog Scale (VAS) for assessment of mental well-being at every visit
6. SDS (Sheehan Disability Scale)
7. Recent and concomitant medications at every visit

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age
2. DSM IV-TR criteria for OCD
3. OCD associated with most distress or most interference in the patient's life as judged by the treating physician
4. Yale-Brown Obsessive Compulsive Scale (YBOCS) total score ≥ 16

Exclusion Criteria:

1. Other primary or co-primary psychiatric disorder which is more distressful for the patient then the OCD, as evaluated by investigator
2. Patients with any history of mania/bipolar disorder
3. Patients using medications which are contraindicated with the use of escitalopram
4. Known contraindication for the use of citalopram or escitalopram.
5. Unable to understand and give informed consent
6. Prominent suicidal ideation (2 points or more in the MADRS "suicidal thoughts" item)
7. Alcohol or substance dependence in the past 6 months
8. Major physical illness
9. Woman currently pregnant or less then 4 weeks after a childbirth, a woman lactating, or a woman of childbearing potential not using a medically accepted form of contraception.
10. Liver function abnormality
11. EKG abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Safety as recorded by adverse-events and side-effects reports.

SECONDARY OUTCOMES:
Reduction in YBOCS scores at week 18

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Barak, MD, MHA, Study Director — Abarbanel MHC
Locations (1):
- Abarbanel MHC, Bat Yam, Israel

REFERENCES:
- [Background] Stengler-Wenzke K, Muller U, Barthel H, Angermeyer MC, Sabri O, Hesse S. Serotonin transporter imaging with [123I]beta-CIT SPECT before and after one year of citalopram treatment of obsessive-compulsive disorder. Neuropsychobiology. 2006;53(1):40-5. doi: 10.1159/000090702. Epub 2006 Jan 4. PMID 16397403
- [Background] Fontenelle LF, Mendlowicz MV, Miguel EC, Versiani M. Citalopram plus reboxetine in treatment-resistant obsessive-compulsive disorder. World J Biol Psychiatry. 2005;6(1):57-9. doi: 10.1080/15622970510029740. PMID 16097406
- [Derived] Rabinowitz I, Baruch Y, Barak Y. High-dose escitalopram for the treatment of obsessive-compulsive disorder. Int Clin Psychopharmacol. 2008 Jan;23(1):49-53. doi: 10.1097/YIC.0b013e3282f0f0c5. PMID 18090508